CLINICAL TRIAL: NCT00723125
Title: Q3week Carboplatin With Weekly Abraxaneä And Avastin + Subsequent Dose-Dense Ac With Avastin As Neoadjuvant Therapy In Resectable And Unresectable (Stage Iia-Iiib) Her2-Negative Breast Cancer
Brief Title: Carboplatin, Abraxane, Avastin as Neoadjuvant Therapy for Her2-Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: William Sikov MD (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor-Investigator, William Sikov MD, Principle Investigator, Brown University
Organization: Brown University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-BR-211A
Record Dates: First submitted 2008-07-15; First posted 2008-07-28 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; Taxes; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Avastin 10 mg/kg IV over 90 minutes day -14
  Abraxane 100 mg/m2 IV over 30 minutes weekly x 12 weeks with Carboplatin at AUC 6 over 30 min IV and Avastin 15 mg/kg IV over 30-90 minutes weeks 1,4,7, and 10
  Avastin 10 mg/kg IV over 30-60 minutes cycles 1-3 (omit dose with cycle 4) Doxorubicin 60 mg/m2* and Cyclophosphamide 600 mg/m2 IV q2weeks x 4 cycles
  Definitive surgery
  Avastin 10 mg/kg IV over 30-60 minutes q2weeks x 34 weeks
  Interventions: Drug: Abraxane; Drug: Carboplatin; Drug: Avastin
- Cohort 2 (Experimental): Abraxane 100 mg/m2 IV over 30 minutes days -14 and -7
  Abraxane 100 mg/m2 IV over 30 minutes weekly x 12 weeks with Carboplatin at AUC 6 over 30 min IV and Avastin 15 mg/kg IV over 30-90 minutes weeks 1,4,7
  Definitive surgery
  Avastin 10 mg/kg IV over 30-60 minutes and Doxorubicin 60 mg/m2* and Cyclophosphamide 600 mg/m2 IV q2weeks x 4 cycles followed by Avastin 10 mg/kg IV over 30-60 minutes q2weeks x 34 weeks OR Avastin 10 mg/kg IV over 30-60 minutes q2weeks x 42 weeks
  Interventions: Drug: Abraxane; Drug: Carboplatin; Drug: Avastin

INTERVENTIONS:
Drug: Abraxane — Abraxane 100 mg/m2 IV over 30 minutes weekly x 12 weeks
  Other Names: Paclitaxel Protein-Bound
Drug: Carboplatin — Carboplatin at AUC 6 over 30 min IV weeks 1,4,7, and 10
  Other Names: Paraplatin
Drug: Avastin — Avastin 15 mg/kg IV over 30-90 minutes weeks 1,4,7, and 10 (in Cohort 2, omit dose of Avastin on week 10)
  Other Names: Bevacizumab

SUMMARY:
In the MDACC/BrUOG neoadjuvant trial with weekly paclitaxel followed by Fluorouracil Plus Doxorubicin and Cyclophosphamide (FAC), the pathologic complete response (pCR) rate in HER2(-) patients was 20%. The investigators' goal is to develop an induction chemotherapy regimen that will have a pCR rate above 30% in patients with HER2(-) disease. Based on a 1-sided 95% confidence interval using normal approximation with an expected pCR rate of at least 35%, approximately 28 patients are required for each cohort. With an assumed pCR rate of at least 35%, the investigators will have approximately 70% statistical power to conclude, with 90% certainty, that the pCR rate with the novel regimen exceeds 20%. The study will accrue approximately 60 patients in two cohorts with an inevaluable rate that does not exceed 10%.

DETAILED DESCRIPTION:
See above brief summary

ELIGIBILITY:
Eligibility criteria

Inclusion criteria:

* Histologically documented adenocarcinoma of the breast
* ANC > 1000 cells
* Female; age > 18
* Zubrod PS 0-1
* Platelets > 100,000
* Stage IIA-IIIB disease
* Total bilirubin < 1.5 ULN
* No evidence of any metastatic disease
* Serum Creatinine < 1.5 gm/dl
* No prior systemic therapy for breast cancer or Creat Cl > 30 ml/min
* Not pregnant or lactating
* Serum ALT < 2.0 ULN
* ER, PR and HER2 status required
* LVEF (MUGA/echo WNL)
* No baseline > 2 neuropathy
* Urine protein: creat ratio < 1.0
* HER2-negative - either IHC 0-1+ or FISH ratio < 2.0
* Hemoglobin > 9 gm/dl
* (FISH testing is required for all HER2 2-3+ tumors by IHC)

Exclusion criteria:

* No Histologically documented adenocarcinoma of the breast
* No-ANC > 1000 cells
* Female; age < 18
* Zubrod PS > 0-1
* Platelets < 100,000
* Stage IV disease
* Total bilirubin > 1.5 ULN
* metastatic disease
* Serum Creatinine > 1.5 gm/dl
* prior systemic therapy for breast cancer or Creat Cl > 30 ml/min
* pregnant or lactating
* Serum ALT > 2.0 ULN baseline > 2 neuropathy
* Urine protein: creat ratio >1.0
* HER2-positive
* Hemoglobin < 9 gm/dl

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2014-05-15 (Actual); Study Completion 2014-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Sikov, MD, Principal Investigator — Brown University
Locations (5):
- United States (5):
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Yale Smilow Cancer Center, New Haven, Connecticut
  - Rhode Island Hsopital, Providence, Rhode Island
  - Women and Infants, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Recruitment Details: DDAC: (dose-dense doxorubicin and cyclophosphamide (DDAC)
Groups:
- Cohort 1: Avastin 10 mg/kg IV over 90 minutes day -14 Abraxane 100 mg/m2 IV over 30 minutes weekly x 12 weeks with Carboplatin at AUC 6 over 30 min IV and Avastin 15 mg/kg IV over 30-90 minutes weeks 1,4,7, and 10 Avastin 10 mg/kg IV over 30-60 minutes cycles 1-3 (omit dose with cycle 4) Doxorubicin 60 mg/m2* and Cyclophosphamide 600 mg/m2 IV q2weeks x 4 cycles Definitive surgery Avastin 10 mg/kg IV over 30-60 minutes q2weeks x 34 weeks
  Cohort 1 and Cohort 2: Abraxane 100 mg/m2 IV over 30 minutes weekly x 12 weeks with Carboplatin at AUC 6 over 30 min IV and Avastin 15 mg/kg IV over 30-90 minutes weeks 1,4,7, and 10 (in Cohort 2, omit dose of Avastin on week 10)
- Cohort 2: Abraxane 100 mg/m2 IV over 30 minutes days -14 and -7 Abraxane 100 mg/m2 IV over 30 minutes weekly x 12 weeks with Carboplatin at AUC 6 over 30 min IV and Avastin 15 mg/kg IV over 30-90 minutes weeks 1,4,7, and 10 (in Cohort 2, omit dose of Avastin on week 10) Definitive surgery Avastin 10 mg/kg IV over 30-60 minutes and Doxorubicin 60 mg/m2* and Cyclophosphamide 600 mg/m2 IV q2weeks x 4 cycles followed by Avastin 10 mg/kg IV over 30-60 minutes q2weeks x 34 weeks OR Avastin 10 mg/kg IV over 30-60 minutes q2weeks x 42 weeks
  Cohort 1 and Cohort 2: Abraxane 100 mg/m2 IV over 30 minutes weekly x 12 weeks with Carboplatin at AUC 6 over 30 min IV and Avastin 15 mg/kg IV over 30-90 minutes weeks 1,4,7, and 10 (in Cohort 2, omit dose of Avastin on week 10)
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 33 (33 pts Neo-adjuvant, 28 evaluable,DDAC: Of 28 pts,27 treated DDAC Avastin:Of 27,15 Avastin post-op) | 27 (27 evaluable Neo-adjuvant Of 27 patients neo-adjuvant, 24 DDAC Of 24 DDAC, 21 Avastin post-op)
Completed | 15 | 21
Not Completed | 18 | 6
Not completed — Met Dx | 1 | 0
Not completed — Withdrawal by Subject | 15 | 6
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 33 | 27 | 60
Age, Continuous [Mean (Full Range); unit: years] | 47.6 [25 to 68] | 45.8 [28 to 63] | 46.8 [25 to 68]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 27 | 59
  >=65 years | 1 | 0 | 1
Sex/Gender, Customized [Number; unit: participants]
  Female | 33 | 27 | 60
Region of Enrollment [Number; unit: participants]
  United States | 33 | 27 | 60

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response Rates at Surgery
Time Frame: at surgery approximately 5 months after initial treatment
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 28 | 27
participants | 16 | 2

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Measure of safety and tolerability according to CTCAE version 3.0
Time Frame: 2 years
Population: Pts with clinical stage IIA-IIIC BrCa
Measure: Number; unit: participants
Groups:
- Cohort 1: Avastin 10 mg/kg IV over 90 minutes day -14
  Abraxane 100 mg/m2 IV over 30 minutes weekly x 12 weeks with Carboplatin at AUC 6 over 30 min IV and Avastin 15 mg/kg IV over 30-90 minutes weeks 1,4,7, and 10
  Avastin 10 mg/kg IV over 30-60 minutes cycles 1-3 (omit dose with cycle 4) Doxorubicin 60 mg/m2* and Cyclophosphamide 600 mg/m2 IV q2weeks x 4 cycles
  Definitive surgery
  Avastin 10 mg/kg IV over 30-60 minutes q2weeks x 34 weeks
  Abraxane: Abraxane 100 mg/m2 IV over 30 minutes weekly x 12 weeks
  Carboplatin: Carboplatin at AUC 6 over 30 min IV weeks 1,4,7, and 10
  Avastin: Avastin 15 mg/kg IV over 30-90 minutes weeks 1,4,7, and 10 (in Cohort 2, omit dose of Avastin on week 10)
- Cohort 2: Abraxane 100 mg/m2 IV over 30 minutes days -14 and -7
  Abraxane 100 mg/m2 IV over 30 minutes weekly x 12 weeks with Carboplatin at AUC 6 over 30 min IV and Avastin 15 mg/kg IV over 30-90 minutes weeks 1,4,7
  Definitive surgery
  Avastin 10 mg/kg IV over 30-60 minutes and Doxorubicin 60 mg/m2* and Cyclophosphamide 600 mg/m2 IV q2weeks x 4 cycles followed by Avastin 10 mg/kg IV over 30-60 minutes q2weeks x 34 weeks OR Avastin 10 mg/kg IV over 30-60 minutes q2weeks x 42 weeks
  Abraxane: Abraxane 100 mg/m2 IV over 30 minutes weekly x 12 weeks
  Carboplatin: Carboplatin at AUC 6 over 30 min IV weeks 1,4,7, and 10
  Avastin: Avastin 15 mg/kg IV over 30-90 minutes weeks 1,4,7, and 10 (in Cohort 2, omit dose of Avastin on week 10)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 28 | 27
participants | 15 | 21

ADVERSE EVENTS:
Time Frame: After run-in therapy neo-adjuvantly, throughout treatment and until completion of follow-up (5 years of follow-up) for a total of approximately 6.5 years
Description: C1 neo: 33 patients enrolled to cohort 1 Neo-adjuvant, only 28 were evaluable C2 neo: 27 enrolled/evaluable cohort 2 Neo-adjuvant C1 DDAC: Of 28 patient evaluable neo-adjuvant, 27 treated DDAC C2 DDAC: Of 27 patients neo-adjuvant, 24 on DDAC C1 Avastin: Of 27 DDAC, 15 Avastin post-op C2 Avastin: Of 24 DDAC, 21 Avastin post-op
Groups:
- Cohort 1 Neo-adjuvant: Avastin 10 mg/kg IV over 90 minutes day -14 Abraxane 100 mg/m2 IV over 30 minutes weekly x 12 weeks with Carboplatin at AUC 6 over 30 min IV and Avastin 15 mg/kg IV over 30-90 minutes weeks 1,4,7, and 10
- Cohort 2 Neo-adjuvant: Abraxane 100 mg/m2 IV over 30 minutes days -14 and -7 Abraxane 100 mg/m2 IV over 30 minutes weekly x 12 weeks with Carboplatin at AUC 6 over 30 min IV and Avastin 15 mg/kg IV over 30-90 minutes weeks 1,4,7, and 10 (in Cohort 2, omit dose of Avastin on week 10)
- Cohort 1 DDAC: Avastin 10 mg/kg IV over 30-60 minutes cycles 1-3 (omit dose with cycle 4) Doxorubicin 60 mg/m2* and Cyclophosphamide 600 mg/m2 IV q2weeks x 4 cycles
- Cohort 2 DDAC: Avastin 10 mg/kg IV over 30-60 minutes and Doxorubicin 60 mg/m2* and Cyclophosphamide 600 mg/m2 IV q2weeks x 4 cycles
- Cohort 1 Adjuvant Post Surgery: Avastin 10 mg/kg IV over 30-60 minutes q2weeks x 34 weeks
- Cohort 2 Adjuvant Post Surgery: Avastin 10 mg/kg IV over 30-60 minutes q2weeks x 34 weeks OR Avastin 10 mg/kg IV over 30-60 minutes q2weeks x 42 weeks
Arm/Group | Cohort 1 Neo-adjuvant | Cohort 2 Neo-adjuvant | Cohort 1 DDAC | Cohort 2 DDAC | Cohort 1 Adjuvant Post Surgery | Cohort 2 Adjuvant Post Surgery
Serious Adverse Events (participants affected / at risk) | 5/28 | 8/27 | 10/27 | 7/24 | 2/15 | 7/21
Other Adverse Events (participants affected / at risk) | 28/28 | 27/27 | 27/27 | 16/24 | 5/15 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Neo-adjuvant (N=28) | Cohort 2 Neo-adjuvant (N=27) | Cohort 1 DDAC (N=27) | Cohort 2 DDAC (N=24) | Cohort 1 Adjuvant Post Surgery (N=15) | Cohort 2 Adjuvant Post Surgery (N=21)
gr 3 Nausea, gr 3 vomiting (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
gr 3 nausea, gr 2 infection with noraml ANC, gr 2 HGB, gr 1 glucose (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
gr 2 non-cardiac chest pain, gr 2 anemia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
gr 3 infection (normal ANC) (cellulitis & pain in buttock - RT infection), gr 1 epistaxis (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
K gr 4,mental status gr 4, ventricular arrythmia gr 4, pneumonia gr 3 (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
gr 2 Pleural effusion (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cr 2, dehydration2, anemia2, weight loss2, fatigue-1, dysgeusia-2, gastritis-2, anorexia-2 (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis gr 3, fever gr 1, fatigue gr 1 (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury gr 2 (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
gr 4 GI Bleed (lesion in colon- villious adenoma) (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FN-gr 1 fever, gr 3 ANC (gr 3 infection) (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FN (fever gr1, ANC 3, infection3)- however during hospitalization ANC rose to grade 4 (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
gr 4 ANC, gr 2 bleeding hemorrhoid, gr 2 rectal pain, dizziness gr 2 (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
left groin abcess- gr 2 1/14/14**amended to grade 3** (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dehydration gr 3, worsening anemia gr 3, diarrhea gr2, anorexia gr 2, ANC 3 (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
gr 3 FN (gr 3 infection, gr 3 ANC), gr 3 mucositis, gr 2 Diarrhea, Gr 2 pain rectal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gr 3 periorbital cellulitis associated with chalazia, gr 2 anemia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gr 4 ANC (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
anemia 2 (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gr 2 dehydration, gr 2 wt loss, gr 2 anorexia, gr 3 esophagitis, gr 2 mucositis, gr 3 ANC, Gr 4 PLT (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gr3 FN, gr3 HGB, Gr2 fatigue, gr2 nausea, gr2 anorexia, gr2 dehydration, gr1 fever, gr1 epistaxis (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — FN-(infection and ANC)
ANC 4, HGB 3, PLT 3 (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
weakness gr 4 (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FN gr 3, ANC 3, anemia gr 2, thrombocytopenia gr 3 (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FN gr3, bradycardia gr1, infection gr3, pancytopenia gr3, sore throat gr1, body aches gr1,rigors gr1 (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — with grade 4 HGB and PLT FN (fever gr 3 and ANC 4)
dehydration2, k3, nausea2, anemia2, cpain2, SOB1, FN, vomiting2, PLT 4, mucositis2, fatigue2 (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — FN - febrile neutropenia :(fever (3) and ANC(4))
gr 2 odynophagia, gr 2 allergic rxn, gr 2 oral thrush, gr 4 ANC (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post Op and Pre-drug- gr 1 fever,gr 2 erythema, gr 2 chills (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post op- wound infection gr 2 on DIEP flap (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FN gr 4 (fever gr 1, ANC 4), cough 2, nasal congestion 2 (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FN (fever gr 1, ANC 4) Anemia 2 (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
bleeding from JP drain grade 1 (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FN- fever gr 1, ANC 4 (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FN gr 3 (fever gr 1, ANC gr 3) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post surgery: gr 3 infection (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
gr 4 skin breakdown (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
gr 2 pleural effusion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
grade 1 fever, gr 3 malignant pleural effusion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
breast cellulitis gr 3, acute renal injury gr 2, diarrhea gr 1, hemmorrhage GI gr 3 (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post Reconstruction Surgery- infection left breast gr 3 (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
post radiation- gr 3 wound complication would dehiscence (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
gr 2 right arm weakness- motor neuropthay, right shoulder pain- r/o TIA (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
secondary malignancy: bladder cancer potentially related to DDAC (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left breast pain gr 2 (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PE gr 4, fever gr 2 (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
post op comp breast cellulitis gr3, migraine gr2 (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Plus:hypocalcemia gr2, hypokalemia gr1, hypomag gr1, anemia gr1, hypophos gr2
related to reconstruction: infection with normal ANC- post complication healing issue (3) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Neo-adjuvant (N=28) | Cohort 2 Neo-adjuvant (N=27) | Cohort 1 DDAC (N=27) | Cohort 2 DDAC (N=24) | Cohort 1 Adjuvant Post Surgery (N=15) | Cohort 2 Adjuvant Post Surgery (N=21)
WBC (Investigations) | 23 (23) | 27 (27) | 5 (5) | 8 (8) | 0 (0) | 3 (3)
ANC (Investigations) | 24 (24) | 22 (22) | 4 (4) | 4 (4) | 0 (0) | 2 (2)
PLT (Investigations) | 25 (25) | 20 (20) | 13 (13) | 2 (2) | 0 (0) | 0 (0)
HGB (Investigations) | 27 (27) | 24 (24) | 21 (21) | 0 (0) | 0 (0) | 0 (0)
Infection (Investigations) | 5 (5) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgias (Investigations) | 0 (0) | 11 (11) | 5 (5) | 0 (0) | 0 (0) | 2 (2)
Creatinine (Investigations) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Investigations) | 4 (4) | 22 (22) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Wt loss (Investigations) | 3 (3) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (Investigations) | 20 (20) | 26 (26) | 17 (17) | 0 (0) | 0 (0) | 4 (4)
Rash (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Investigations) | 12 (12) | 22 (22) | 11 (11) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Investigations) | 6 (6) | 9 (9) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Mucositis (Investigations) | 6 (6) | 16 (16) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Investigations) | 5 (5) | 16 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Investigations) | 9 (9) | 14 (14) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
LFTs (Investigations) | 10 (10) | 12 (12) | 7 (7) | 0 (0) | 0 (0) | 3 (3)
Neurosensory (Investigations) | 3 (3) | 17 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuromuscular (Investigations) | 4 (4) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Investigations) | 4 (4) | 5 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Investigations) | 5 (5) | 7 (7) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesmia (Investigations) | 12 (12) | 4 (4) | 10 (10) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Investigations) | 5 (5) | 12 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alk-Phos abnormality (Investigations) | 4 (4) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cough (Investigations) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
epistaxis or bleeding (Investigations) | 13 (13) | 24 (24) | 5 (5) | 12 (12) | 2 (2) | 7 (7)
Chest Pain/Bradycardia (Investigations) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
HTN (Investigations) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 7 (7)
SOB (Investigations) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ocular (Investigations) | 0 (0) | 13 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbili (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No